CLINICAL TRIAL: NCT00359645
Title: DEPISTORL - THANCS (Trial of Head And Neck Cancer Screening) Randomized Multicenter Trial to Assess the Impact of a Screening Program for Heavy Alcohol Drinkers and Smokers Treated in Alcohol Addiction Clinics on Upper Aerodigestive Tract Cancer Mortality.
Brief Title: Randomized Trial to Assess the Impact of a Screening Program on Upper Aerodigestive Tract Cancer Mortality in a High Risk Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEPISTORL - THANCS; CET 1172
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pharynx Cancer; Larynx Cancer; Oral Cavity Cancer; Oesophageal Cancer
Keywords: Screening; Upper aerodigestive tract cancer; Alcohol; Tobacco; Randomized trial
MeSH Terms: conditions — Pharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Esophageal Neoplasms

ARMS (2):
- Control (No Intervention): Annual auto questionnaire
- Screening (Experimental): Annual screening of Head and Neck cancer
  Interventions: Procedure: Screening by head and neck clinical examination with a fiberoptic nasolaryngoscopy and an oesopharyngeal brush biopsy annually during 3 years

INTERVENTIONS:
Procedure: Screening by head and neck clinical examination with a fiberoptic nasolaryngoscopy and an oesopharyngeal brush biopsy annually during 3 years
  Arms: Screening

SUMMARY:
Randomized multicenter trial to assess the impact of a screening program for heavy alcohol drinkers and smokers treated in alcohol addiction clinics on upper aerodigestive tract cancer mortality.

DETAILED DESCRIPTION:
Upper aerodigestive tract (UADT) carcinomas (oral cavity and pharynx (63%), larynx (17%) and esophagus (20%)), are frequent in France with 25.000 new cases annually estimated in 2000, representing 13% of men cancer (3rd rank). Five-year specific survival rate is approximately 50% (11.000 deaths per year) and has not improved in over three decades, primarily due to the advanced stage at presentation. UADT cancers are also associated with profound disease- and treatment-related morbidity, with alterations in speech and feeding functions, aesthetic disability, with familial and social consequences.

The high-risk population is well characterized. A synergistic effect of tobacco smoking and alcohol drinking increases the risk of developing a carcinoma by more than 100 fold. Each year, 30.000 alcohol drinkers are treated in alcohol addiction clinics and could benefit from cancer detection. Nonrandomized pilot studies have showed that a UADT cancers screening trial could be undertaken in these clinics.

Study design: prospective randomized trial comparing an observation group and a screening group. Subjects in the screening group will undergo annual screening test including head and neck clinical examination with a fiberoptic nasolaryngoscopy and an oesopharyngeal brush biopsy with cytological examination during a 3-years period. In case of a positive test, patients will undergo head and neck panendoscopy and/or digestive flexible endoscopy and/or biopsy. After the screening period, subjects will be followed during 2 additional years by annual health questionnaires. Subjects of the observation group will be followed during 5 years by annual health questionnaires. Recruitment will be performed in alcohol addiction clinics and screening tests and confirmation exams in the closest specialized head and neck clinics.

The primary objective is to demonstrate a decrease in the UADT cancer mortality after a screening strategy, including head and neck clinical examination with a fiberoptic nasolaryngoscopy and an oesopharyngeal brush biopsy with cytological examination repeated annually during 3 years. Subjects will be followed during 5 years. A sample size of 10.000 subjects in each group allows the detection of a 33% reduction in the specific mortality rate, with a power of 80% and with a one sided a-risk of 5%.

ELIGIBILITY:
Inclusion Criteria:

* current or previous heavy smokers (smoked >= 20 years) and alcohol drinkers who need specialized care

Exclusion Criteria:

* Head and neck clinical examination during the past 6 months
* History of squamous cell carcinoma of the upper aero-digestive tract.
* Recent digestive hemorrhage from varicose esophagus

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1993 (Actual)
Dates: Start 2006-06-21 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Upper aerodigestive tract cancer mortality | 5 years

SECONDARY OUTCOMES:
Screening test morbidity | 1 week
Upper aerodigestive tract cancer incidence | 5 years
Upper aerodigestive tract cancer stage | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane TEMAM, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (35):
- France (35):
  - Centre Hospitalier MONTPERRIN, Aix-en-Provence
  - CHIAB Annemasse Bonneville, Annemasse
  - Centre Hospitalier d'ARRAS, Arras
  - CHS de L'Yonne, Auxerre
  - Chg Beziers, Béziers
  - C.A.S.A., Clermont
  - CHU Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier de DIEPPE, Dieppe
  - CHU le Bocage, Dijon
  - Centre Hospitalier Louis Sevestre, La Membrolle-sur-Choisille
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier de LENS, Lens
  - CHU de Lille, Lille
  - CHBS Lorient, Lorient
  - Centre hospitalier Lyon sud, Lyon
  - Centre Hospitalier des Chanaux, Mâcon
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital ARCHET II, Nice
  - Centre ANPAA d'Orléans, Orléans
  - Centre Paul Cézanne, Orléans
  - Hôpital de la Source, Orléans
  - Clinique Philae, Pont-Péan
  - Centre Hospitalier du Centre Bretagne, Pontivy
  - Centre ANPAA 51 de Reims, Reims
  - CHU Hôpital Pontchaillou, Rennes
  - Hopital de Saint Cloud, Saint-Cloud
  - CHR de la Réunion, Saint-denis de La Reunion
  - Ch Saint-Egreve, Saint-Égrève
  - Centre de soins de suite Marienbronn, Soultz-sous-Forêts
  - CHU de Strasbourg - Hôpital Hautepierre, Strasbourg
  - Hôpitaux du Leman, Thonon-les-Bains
  - Chba Vannes, Vannes
  - Hopital Paul Brousse, Villejuif
  - Institut_Gustave-Roussy, Villejuif

REFERENCES:
- See also: DepistORL — http://www.depistorl.org